CLINICAL TRIAL: NCT02948959
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Evaluate the Efficacy and Safety of Dupilumab in Children 6 to <12 Years of Age With Uncontrolled Persistent Asthma
Brief Title: Evaluation of Dupilumab in Children With Uncontrolled Asthma
Acronym: VOYAGE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EFC14153; 2016-001607-23 (EudraCT Number); U1111-1179-4851 (Other: UTN)
Record Dates: First submitted 2016-10-27; First posted 2016-10-31 (Estimated); Results first posted 2021-10-20 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo (for Dupilumab), subcutaneous (SC) injection every 2 weeks (q2w) for 52 weeks in combination with stable-dose background therapy of medium-dose inhaled corticosteroids (ICS) with a second controller medication (i.e., long-acting β2 agonist [LABA], long acting muscarinic antagonist [LAMA], leukotriene receptor antagonist [LTRA] or methylxanthines) or high-dose ICS alone or high-dose ICS with second controller medication. Albuterol/salbutamol or levalbuterol/levosalbutamol was given as reliever medication. Participants were followed up for 12 weeks after last dose (i.e. up to Week 64).
  Interventions: Drug: Placebo; Drug: Asthma Controller Therapies; Drug: Asthma Reliever Therapies
- Dupilumab (Experimental): Dupilumab 200 milligrams (mg) (in 1.14 milliliters [mL] for >30 kilograms [kg] bodyweight [BW]) or 100 mg (in 0.67 mL for less than or equal to (<=) 30 kg BW), SC injection q2w for 52 weeks in combination with stable-dose background therapy of medium-dose ICS with a second controller medication (i.e., LABA, LAMA, LTRA] or methylxanthines) or high-dose ICS alone or high-dose ICS with second controller medication. Albuterol/salbutamol or levalbuterol/levosalbutamol was given as reliever medication. Participants were followed up for 12 weeks after last dose (i.e. up to Week 64).
  Interventions: Drug: Dupilumab; Drug: Asthma Controller Therapies; Drug: Asthma Reliever Therapies

INTERVENTIONS:
Drug: Dupilumab — Pharmaceutical form: Solution
  Route of administration: Subcutaneous
  Other Names: SAR231893 (REGN668)
  Arms: Dupilumab
Drug: Placebo — Pharmaceutical form: Solution
  Route of administration: Subcutaneous
  Arms: Placebo
Drug: Asthma Controller Therapies — Pharmaceutical form: Aerosol, capsules, tablets, oral solution
  Route of administration: Inhaled, oral
Drug: Asthma Reliever Therapies — Pharmaceutical form: Nebulized, aerosol
  Route of administration: Inhaled

SUMMARY:
Primary Objective:

To evaluate the efficacy of dupilumab in children 6 to less than (<) 12 years of age with uncontrolled persistent asthma.

Secondary Objective:

To evaluate in children 6 to <12 years of age with uncontrolled persistent asthma:

* The safety and tolerability of dupilumab.
* The evaluate the effect of dupilumab in improving participant reported outcomes including health related quality of life.
* The dupilumab systemic exposure and incidence of anti-drug antibodies.
* The evaluate the association between dupilumab treatment and pediatric immune responses to vaccines: any vaccination for tetanus, diphtheria, pertussis and/or seasonal trivalent/quadrivalent influenza vaccine.

DETAILED DESCRIPTION:
The total study duration per participant was up to 69 weeks, consisted of a screening period of 3-5 weeks, a randomized treatment period of 52 weeks and a post-treatment period of 12 weeks.

ELIGIBILITY:
Inclusion criteria :

Children 6 to <12 years of age, with a physician diagnosis of persistent asthma for greater than or equal to (>=)12 months prior to screening, based on clinical history and examination, pulmonary function parameters according to Global initiative for asthma (GINA) 2015 Guidelines and the following criteria:

* Existing background therapy of medium-dose ICS with second controller medication (i.e., long-acting β2 agonist , leukotriene receptor antagonist, long acting muscarinic antagonist, or methylxanthines) or high-dose ICS alone or high-dose ICS with second controller, for at least 3 months with a stable dose >=1 month prior to Screening Visit 1.
* Pre-bronchodilator forced expiratory volume in 1 second (FEV1) <=95 percentage (%) of predicted normal or pre bronchodilator FEV1/forced vital capacity ratio <0.85 at Screening and Baseline Visits.
* Reversibility of at least 10% in FEV1 after the administration of 200 to 400 micrograms (mcg; 2 to 4 puff inhalations with metered-dose inhaler [MDI]) of albuterol/salbutamol or 45 to 90 mcg (2 to 4 puffs with MDI) of levalbuterol/levosalbutamol reliever medication before randomization (up to 3 opportunities during the same visit were allowed with a maximum of 12 puffs of reliever medication if tolerated by the participant).
* Must had experienced, within 1 year prior to Screening Visit 1, any of the following events:

  * Treatment with a systemic corticosteroid (oral or parenteral), as prescribed by a healthcare professional for worsening asthma at least once or,
  * Hospitalization or emergency visit for worsening asthma.
* Evidence of uncontrolled asthma, with at least one of the following criteria during the 4 (±1) weeks Screening Period:

  * Asthma Control Questionnaire-Interviewer Administered (ACQ-IA) ACQ-5 score >=1.5 on at least one day of the Screening Period.
  * Use of reliever medication (i.e., albuterol/salbutamol or levalbuterol/levosalbutamol), other than as a preventive for exercise induced bronchospasm, on 3 or more days per week, in at least one week during the Screening Period.
  * Sleep awakening due to asthma symptoms requiring use of reliever medication at least once during the Screening Period.
  * Asthma symptoms 3 or more days per week in at least one week during the Screening Period.

Exclusion criteria:

* Participants <6 or >=12 years of age.
* Participants with <16 kg bodyweight.
* Any other chronic lung disease (cystic fibrosis, bronchopulmonary dysplasia, etc.), which may impair lung function.
* A participant with any history of life threatening asthma (ie, extreme exacerbation that requires intubation).
* Co-morbid disease that might interfere with the evaluation of investigational medicinal product.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 408 (Actual)
Dates: Start 2017-04-21 (Actual); Primary Completion 2020-08-26 (Actual); Study Completion 2020-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (99):
- United States (18):
  - Investigational Site Number 840031, Birmingham, Alabama
  - Investigational Site Number 840002, Gilbert, Arizona
  - Investigational Site Number 840012, Tucson, Arizona
  - Investigational Site Number 840001, Rolling Hills Estates, California
  - Investigational Site Number 840036, Owensboro, Kentucky
  - Investigational Site Number 840016, Ann Arbor, Michigan
  - Investigational Site Number 840006, St Louis, Missouri
  - Investigational Site Number 840022, Lincoln, Nebraska
  - Investigational Site Number 840023, Great Neck, New York
  - Investigational Site Number 840035, New York, New York
  - Investigational Site Number 840013, New York, New York
  - Investigational Site Number 840007, Rochester, New York
  - Investigational Site Number 840004, Charlotte, North Carolina
  - Investigational Site Number 840021, Durham, North Carolina
  - Investigational Site Number 840008, Cincinnati, Ohio
  - Investigational Site Number 840024, Edmond, Oklahoma
  - Investigational Site Number 840003, San Antonio, Texas
  - Investigational Site Number 840018, La Crosse, Wisconsin
- Argentina (5):
  - Investigational Site Number 032004, Buenos Aires
  - Investigational Site Number 032003, Buenos Aires
  - Investigational Site Number 032002, Caba
  - Investigational Site Number 032001, Caba
  - Investigational Site Number 032006, Mendoza
- Australia (4):
  - Investigational Site Number 036001, Campbelltown
  - Investigational Site Number 036005, North Adelaide
  - Investigational Site Number 036003, Parkville/Melbourne
  - Investigational Site Number 036002, South Brisbane
- Brazil (7):
  - Investigational Site Number 076008, Blumenau
  - Investigational Site Number 076001, Porto Alegre
  - Investigational Site Number 076007, Porto Alegre
  - Investigational Site Number 076003, São Paulo
  - Investigational Site Number 076002, São Paulo
  - Investigational Site Number 076004, São Paulo
  - Investigational Site Number 076006, Sorocaba
- Canada (4):
  - Investigational Site Number 124004, Edmonton
  - Investigational Site Number 124002, Hamilton
  - Investigational Site Number 124001, Montreal
  - Investigational Site Number 124003, Québec
- Chile (6):
  - Investigational Site Number 152003, Santiago
  - Investigational Site Number 152005, Santiago
  - Investigational Site Number 152009, Santiago
  - Investigational Site Number 152001, Valdivia
  - Investigational Site Number 152007, Viña del Mar
  - Investigational Site Number 152002, Viña del Mar
- Colombia (2):
  - Investigational Site Number 170004, Antioquia
  - Investigational Site Number 170002, Cali
- Hungary (8):
  - Investigational Site Number 348006, Budapest
  - Investigational Site Number 348002, Gyula
  - Investigational Site Number 348012, Mezőkövesd
  - Investigational Site Number 348005, Szeged
  - Investigational Site Number 348001, Székesfehérvár
  - Investigational Site Number 348008, Szigetvár
  - Investigational Site Number 348003, Töröbálint
  - Investigational Site Number 348007, Zalaegerszeg
- Italy (5):
  - Investigational Site Number 380007, Catania
  - Investigational Site Number 380003, Florence
  - Investigational Site Number 380004, Padua
  - Investigational Site Number 380005, Roma
  - Investigational Site Number 380001, Verona
- Lithuania (5):
  - Investigational Site Number 440002, Kaunas
  - Investigational Site Number 440005, Šiauliai
  - Investigational Site Number 440003, Utena
  - Investigational Site Number 440001, Vilnius
  - Investigational Site Number 440004, Vilnius
- Mexico (5):
  - Investigational Site Number 484006, Chihuahua City
  - Investigational Site Number 484004, Chihuahua City
  - Investigational Site Number 484003, Durango
  - Investigational Site Number 484001, Monterrey
  - Investigational Site Number 484002, Veracruz
- Poland (2):
  - Investigational Site Number 616001, Lodz
  - Investigational Site Number 616002, Poznan
- Investigational Site Number 642001, Bucharest, Romania
- Russia (6):
  - Investigational Site Number 643006, Moscow
  - Investigational Site Number 643004, Perm
  - Investigational Site Number 643005, Saint Petersburg
  - Investigational Site Number 643002, Saint Petersburg
  - Investigational Site Number 643001, Saint Petersburg
  - Investigational Site Number 643003, Saint Petersburg
- South Africa (2):
  - Investigational Site Number 710004, Cape Town
  - Investigational Site Number 710001, Cape Town
- Spain (5):
  - Investigational Site Number 724001, Barcelona
  - Investigational Site Number 724006, Esplugues de Llobregat
  - Investigational Site Number 724005, Pozuelo de Alarcón
  - Investigational Site Number 724002, Santiago de Compostela
  - Investigational Site Number 724003, Valencia
- Turkey (Türkiye) (6):
  - Investigational Site Number 792005, Adana
  - Investigational Site Number 792008, Ankara
  - Investigational Site Number 792001, Ankara
  - Investigational Site Number 792006, Bursa
  - Investigational Site Number 792003, Istanbul
  - Investigational Site Number 792004, Istanbul
- Ukraine (8):
  - Investigational Site Number 804007, Chernivtsi
  - Investigational Site Number 804004, Dnipro
  - Investigational Site Number 804011, Ivano-Frankivsk
  - Investigational Site Number 804005, Kharkiv
  - Investigational Site Number 804008, Kryvyi Rig
  - Investigational Site Number 804001, Kyiv
  - Investigational Site Number 804002, Zaporizhzhya
  - Investigational Site Number 804003, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Jackson DJ, Hamelmann E, Roberts G, Bacharier LB, Xia C, Gall R, Ledanois O, Coleman A, Tawo K, Jacob-Nara JA, Radwan A, Rowe PJ, Deniz Y. Dupilumab Efficacy and Safety in Children With Moderate to Severe Asthma and High Blood Eosinophils: A Post Hoc Analysis of VOYAGE. J Allergy Clin Immunol Pract. 2025 Mar;13(3):568-575. doi: 10.1016/j.jaip.2024.11.014. Epub 2024 Nov 28. PMID 39613097
- [Derived] Guilbert TW, Murphy KR, Hamelmann E, Ross KR, Gupta A, Fiocchi A, Xia C, Gall R, Ledanois O, Radwan A, Jacob-Nara JA, Rowe PJ, Deniz Y. Impact of Lung Function on Asthma Exacerbation Rates in Children Treated with Dupilumab: The VOYAGE Study. J Asthma Allergy. 2024 Feb 8;17:81-87. doi: 10.2147/JAA.S425101. eCollection 2024. PMID 38347908
- [Derived] Bacharier LB, Pavord ID, Maspero JF, Jackson DJ, Fiocchi AG, Mao X, Jacob-Nara JA, Deniz Y, Laws E, Mannent LP, Amin N, Akinlade B, Staudinger HW, Lederer DJ, Hardin M. Blood eosinophils and fractional exhaled nitric oxide are prognostic and predictive biomarkers in childhood asthma. J Allergy Clin Immunol. 2024 Jul;154(1):101-110. doi: 10.1016/j.jaci.2023.09.044. Epub 2024 Jan 23. PMID 38272375
- [Derived] Bacharier LB, Guilbert TW, Katelaris CH, Deschildre A, Phipatanakul W, Liu D, Altincatal A, Mannent LP, Amin N, Laws E, Akinlade B, Jacob-Nara JA, Deniz Y, Rowe PJ, Lederer DJ, Hardin M. Dupilumab Improves Lung Function Parameters in Pediatric Type 2 Asthma: VOYAGE Study. J Allergy Clin Immunol Pract. 2024 Apr;12(4):948-959. doi: 10.1016/j.jaip.2023.12.006. Epub 2023 Dec 11. PMID 38092225
- [Derived] Fiocchi AG, Phipatanakul W, Zeiger RS, Durrani SR, Cole J, Msihid J, Gall R, Jacob-Nara JA, Deniz Y, Rowe PJ, Lederer DJ, Hardin M, Zhang Y, Khan AH. Dupilumab leads to better-controlled asthma and quality of life in children: the VOYAGE study. Eur Respir J. 2023 Nov 2;62(5):2300558. doi: 10.1183/13993003.00558-2023. Print 2023 Nov. PMID 37734856
- [Derived] Papadopoulos NG, Szefler SJ, Bacharier LB, Maspero JF, Domingo C, Fiocchi A, Lee JK, Daizadeh N, Lederer DJ, Hardin M, Gall R, Djandji M, Siddiqui S, Jacob-Nara JA, Deniz Y, Rowe PJ. Assessment of dupilumab in children with moderate-to-severe type 2 asthma with or without evidence of allergic asthma. Allergy. 2023 Aug;78(8):2157-2167. doi: 10.1111/all.15743. Epub 2023 May 25. PMID 37059696
- [Derived] Jackson DJ, Bacharier LB, Phipatanakul W, Sher L, Domingo C, Papadopoulos N, Modena B, Li N, Xia C, Kamal MA, Dillon M, Wolfe K, Gall R, Amin N, Mannent LP, Laws E, Rowe PJ, Jacob-Nara JA, Deniz Y, Lederer DJ, Hardin M, Xu C. Dupilumab pharmacokinetics and effect on type 2 biomarkers in children with moderate-to-severe asthma. Ann Allergy Asthma Immunol. 2023 Jul;131(1):44-51.e4. doi: 10.1016/j.anai.2023.03.014. Epub 2023 Mar 22. PMID 36958470
- [Derived] Bacharier LB, Maspero JF, Katelaris CH, Fiocchi AG, Gagnon R, de Mir I, Jain N, Sher LD, Mao X, Liu D, Zhang Y, Khan AH, Kapoor U, Khokhar FA, Rowe PJ, Deniz Y, Ruddy M, Laws E, Patel N, Weinreich DM, Yancopoulos GD, Amin N, Mannent LP, Lederer DJ, Hardin M; Liberty Asthma VOYAGE Investigators. Dupilumab in Children with Uncontrolled Moderate-to-Severe Asthma. N Engl J Med. 2021 Dec 9;385(24):2230-2240. doi: 10.1056/NEJMoa2106567. PMID 34879449

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 90 active centers in 17 countries. A total of 631 participants were screened between 21 April 2017 and 22 July 2019, of which 408 participants were enrolled and randomized to receive dupilumab or placebo. A total of 223 participants failed screening mainly due to failure to meet inclusion criteria.
Pre-assignment Details: Randomization was stratified by inhaled corticosteroids (ICS) dose level (medium or high), blood eosinophils count (less than [<] 300 cells per microliter and greater than or equal to [>=] 300 cells per microliter), and region (Latin America, Eastern Europe, and Western countries). Treatment assignment was done by Interactive Voice/Web Response System (2:1 ratio) to receive dupilumab or placebo.
Groups:
- Placebo: Placebo (for Dupilumab), subcutaneous (SC) injection every 2 weeks (q2w) for 52 weeks in combination with stable-dose background therapy of medium-dose ICS with a second controller medication (i.e., long-acting β2 agonist [LABA], long acting muscarinic antagonist [LAMA], leukotriene receptor antagonist [LTRA] or methylxanthines) or high-dose ICS alone or high-dose ICS with second controller medication. Albuterol/salbutamol or levalbuterol/levosalbutamol was given as reliever medication. Participants were followed up for 12 weeks after last dose (i.e. up to Week 64).
- Dupilumab: Dupilumab 200 milligrams (mg) (in 1.14 milliliters [mL] for >30 kilograms (kg) bodyweight [BW]) or 100 mg (in 0.67 mL for <=30 kg BW), SC injection q2w for 52 weeks in combination with stable-dose background therapy of medium-dose ICS with a second controller medication (i.e., LABA, LAMA, LTRA or methylxanthines) or high-dose ICS alone or high-dose ICS with second controller medication. Albuterol/salbutamol or levalbuterol/levosalbutamol was given as reliever medication. Participants were followed up for 12 weeks after last dose (i.e. up to Week 64).
Period: 52 Weeks Treatment Period
Arm/Group | Placebo | Dupilumab
Started (Randomized.) | 135 | 273
Treated | 135 | 270
Safety Population (Participants who actually received at least 1 dose or part of a dose of investigational medicinal product (IMP), analyzed according to the treatment actually received.) | 134 (1 participant randomized to placebo received dupilumab; counted in dupilumab arm for safety analysis.) | 271 (1 participant randomized to placebo received dupilumab; counted in dupilumab arm for safety analysis.)
Type 2 Inflammatory Asthma Phenotype Population (Randomized participants with baseline blood eosinophils >=150 cells per microliter or baseline fractional exhaled nitric oxide (FeNO) >=20 parts per billion (ppb).) | 114 | 236
Baseline Blood Eosinophils Count >=300 Cells Per Microlitre Population (Randomized participants with baseline blood eosinophil count >=300 cells per microliter.) | 84 | 175
Completed | 130 | 248
Not Completed | 5 | 25
Not completed — Poor compliance to protocol | 0 | 2
Not completed — Adverse Event | 2 | 5
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Participant used protocol prohibited vaccine | 1 | 6
Not completed — Randomized by error | 0 | 5
Not completed — Randomized and not treated | 0 | 3
Not completed — Non-compliant to study treatment | 0 | 1
Not completed — Change of residence location | 0 | 1
Period: 12 Weeks Follow-up Period
Arm/Group | Placebo | Dupilumab
Started (Only participants who completed treatment, did not continue to 1-year long-term open-label extension study (LTS14424; NCT03560466) entered Period 2 (12-week posttreatment follow-up period).) | 9 | 31
Completed | 4 | 19
Not Completed | 5 | 12
Not completed — Adverse Event | 0 | 2
Not completed — Poor compliance to protocol | 1 | 2
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Randomized by error | 0 | 3
Not completed — Change of residence location | 0 | 2
Not completed — Study site closure | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on intent to treat population which included all randomized participants.
Groups:
- Placebo: Placebo (for Dupilumab), SC injection q2w for 52 weeks in combination with stable-dose background therapy of medium-dose ICS with a second controller medication (i.e., LABA, LAMA, LTRA or methylxanthines) or high-dose ICS alone or high-dose ICS with second controller medication. Albuterol/salbutamol or levalbuterol/levosalbutamol was given as reliever medication. Participants were followed up for 12 weeks after last dose (i.e. up to Week 64).
- Dupilumab: Dupilumab 200 mg (in 1.14 mL for >30 kg BW) or 100 mg (in 0.67 mL for <=30 kg BW), SC injection q2w for 52 weeks in combination with stable-dose background therapy of medium-dose ICS with a second controller medication (i.e., LABA, LAMA, LTRA or methylxanthines) or high-dose ICS alone or high-dose ICS with second controller medication. Albuterol/salbutamol or levalbuterol/levosalbutamol was given as reliever medication. Participants were followed up for 12 weeks after last dose (i.e. up to Week 64).
- Total: Total of all reporting groups
Arm/Group | Placebo | Dupilumab | Total
Number analyzed (Participants) | 135 | 273 | 408
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.9 (1.6) | 8.9 (1.7) | 8.9 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 98 | 146
  Male | 87 | 175 | 262
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian/White | 118 | 242 | 360
  Black/of African descent | 9 | 11 | 20
  Asian/Oriental | 0 | 2 | 2
  American Indian or Alaska Native | 0 | 1 | 1
  Other | 8 | 17 | 25

OUTCOME MEASURES:

1. Primary Outcome: Annualized Rate of Severe Exacerbation Events During the 52-Week Treatment Period: Baseline Blood Eosinophils >=300 Cells Per Microliter Population
Description: A severe asthma exacerbation event was defined as a deterioration of asthma during the 52-week treatment period requiring: use of systemic corticosteroids for >=3 days; and/or hospitalization or emergency room visit because of asthma requiring systemic corticosteroid treatment. Annualized event rate was defined as the total number of severe exacerbation events that occurred during the 52-week treatment period divided by the total number of participant-years followed in the 52-week treatment period.
Time Frame: Baseline to Week 52
Population: Analysis was performed on baseline blood eosinophils >=300 cells per microliter population which included the randomized participants with baseline blood eosinophil count >=300 cells per microliter.
Measure: Number (95% Confidence Interval); unit: exacerbations per participant-years
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 84 | 175
exacerbations per participant-years | 0.665 [0.467 to 0.949] | 0.235 [0.160 to 0.345]
Statistical Analysis 1: Comparison: Placebo vs Dupilumab; Risk ratio and p-value was derived using negative binomial model with total number of events onset from randomization up to Week 52 visit or last contact date (whichever comes earlier) as response variable, with treatment group, age, baseline weight group, region, baseline eosinophil level, baseline FeNO level, baseline ICS dose level and number of severe exacerbation events within 1 year prior to study as covariates and log-transformed standardized observation duration as an offset variable; Test type: Superiority — To control the type-I error rate for the analysis of outcome measure, a hierarchical testing procedure was applied at a 2-sided 5% significant level. Testing was then performed sequentially in the order endpoints were reported. Hierarchical testing sequence continued only if the previous endpoint was statistically significant; p < 0.0001, Negative binomial model — Threshold for statistical significance at 5% significant level; Risk Ratio (RR) = 0.353, 95% CI 2-sided [0.222 to 0.562] — Risk ratio, also called relative risk compares the risk (rate) of an event among one group with the risk (rate) among another group

2. Primary Outcome: Annualized Rate of Severe Exacerbation Events During the 52-Week Treatment Period: Type 2 Inflammatory Asthma Phenotype Population
Description: as for outcome 1
Time Frame: Baseline to Week 52
Population: Analysis was performed on type 2 inflammatory asthma phenotype population which included the randomized participants with baseline blood eosinophil count >=150 cells per microliter or baseline FeNO >=20 ppb.
Measure: Number (95% Confidence Interval); unit: exacerbations per participant-years
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 114 | 236
exacerbations per participant-years | 0.748 [0.542 to 1.034] | 0.305 [0.223 to 0.416]
Statistical Analysis 1: Comparison: Placebo vs Dupilumab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — Testing was performed according to the hierarchical testing procedure (continued only if the previous endpoint was statistically significant); p < 0.0001, Negative binomial model — Threshold for statistical significance at 5% significant level; Risk Ratio (RR) = 0.407, 95% CI 2-sided [0.274 to 0.605] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline in Pre-bronchodilator Percent Predicted Forced Expiratory Volume in 1 (FEV1) Second at Week 12: Baseline Blood Eosinophils >=300 Cells Per Microliter Population
Description: FEV1 was the volume of air (in liters) exhaled from the lungs in the first second of a forced expiration as measured by spirometer. LS means and SE were derived from MMRM model with change from baseline in pre-bronchodilator % predicted FEV1 value up to Week 12 as the response variable, and treatment, baseline weight group, region, ethnicity, baseline eosinophil level, baseline FeNO level, baseline ICS dose level, visit, treatment by-visit interaction, baseline % predicted FEV1 value and baseline-by-visit interaction as covariates.
Time Frame: Baseline, Week 12
Population: Analysis was performed on baseline blood eosinophils >=300 cells per microliter population. Here, 'Overall number of participants analyzed'=participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: percent predicted FEV1
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 80 | 168
percent predicted FEV1 | 4.83 (1.54) | 10.15 (1.12)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab; P-value and LS mean difference were derived from MMRM model with change from baseline in pre-bronchodilator % predicted FEV1 value up to Week 12 as the response variable, and treatment, baseline weight group, region, ethnicity, baseline eosinophil level, baseline FeNO level, baseline ICS dose level, visit, treatment by-visit interaction, baseline % predicted FEV1 value and baseline-by-visit interaction as covariates; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.0036, Mixed-effect model with repeated measure — Threshold for statistical significance at 5% significant level; LS mean difference = 5.32, 95% CI 2-sided [1.76 to 8.88]

4. Secondary Outcome: Change From Baseline in Pre-bronchodilator Percent Predicted Forced Expiratory Volume in 1 Second (FEV1) at Week 12: Type 2 Inflammatory Asthma Phenotype Population
Description: FEV1 was the volume of air (in liters) exhaled from the lungs in the first second of a forced expiration as measured by spirometer. Least square (LS) means and standard error (SE) were derived from mixed-effect model with repeated measures (MMRM) model with change from baseline in pre-bronchodilator % predicted FEV1 value up to Week 12 as the response variable, and treatment, baseline weight group, region, ethnicity, baseline eosinophil level, baseline FeNO level, baseline ICS dose level, visit, treatment by-visit interaction, baseline % predicted FEV1 value and baseline-by-visit interaction as covariates.
Time Frame: Baseline, Week 12
Population: Analysis was performed on type 2 inflammatory asthma phenotype population. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: percent predicted FEV1
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 110 | 229
percent predicted FEV1 | 5.32 (1.36) | 10.53 (1.01)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab; P-value and LS mean difference were derived from MMRM model with change from baseline in pre-bronchodilator % predicted FEV1 value up to Week 12 as the response variable, and treatment, baseline weight group, region, ethnicity, baseline eosinophil level, baseline FeNO level, baseline ICS dose level, visit, treatment by-visit interaction, baseline % predicted FEV1 value and baseline-by visit interaction as covariates; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.0009, Mixed-effect model with repeated measure — Threshold for statistical significance at 5% significant level; LS mean difference = 5.21, 95% CI 2-sided [2.14 to 8.27]

5. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire-Interviewer Administered, 7-question Version (ACQ-7-IA) at Week 24: Baseline Blood Eosinophils >=300 Cells Per Microliter Population
Description: ACQ-7-IA had 7 questions, which assessed: frequency of nocturnal awakenings, severity of asthma symptoms in the mornings, limitation of daily activities, shortness of breath due to asthma and wheeze, reliever medication use, and FEV1 (% predicted). Participants recalled their previous week asthma and answered 5 symptom questions on 7-point scale ranging from 0 (no impairment) to 6 (maximum impairment). Total score: mean of scores of all 7 questions; ranging from 0 (totally controlled) to 6 (severely uncontrolled), higher score indicated lower asthma control. LS means and SE were derived from MMRM model with change from baseline in ACQ-7-IA values up to Week 52 as response variable and treatment, age, baseline weight group, region, baseline eosinophil level, baseline FeNO level, baseline ICS dose level, visit, treatment by-visit interaction, baseline ACQ-7-IA value and baseline-by-visit interaction as covariates.
Time Frame: Baseline, Week 24
Population: Analysis was performed on baseline blood eosinophils >=300 cells per microliter population. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 80 | 166
score on a scale | -0.88 (0.09) | -1.34 (0.06)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab; P-value and LS mean difference were derived from MMRM model with change from baseline in ACQ-7-IA up to Week 52 as the response variable, and treatment, age, weight group, region, baseline eosinophil level, baseline FeNO level, baseline ICS dose level, visit, treatment by-visit interaction, baseline ACQ-7-IA and baseline-by-visit interaction as covariates; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.0001, Mixed-effect model with repeated measure — Threshold for statistical significance at 5% significant level; LS mean difference = -0.46, 95% CI 2-sided [-0.66 to -0.26]

6. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire-Interviewer Administered, 7-question Version at Week 24: Type 2 Inflammatory Asthma Phenotype Population
Description: ACQ-7-IA had 7 questions, which assessed: frequency of nocturnal awakenings, severity of asthma symptoms in the mornings, limitation of daily activities due to asthma, shortness of breath due to asthma and wheeze, reliever medication use, and FEV1 (% predicted). Participants recalled their previous week asthma and answered 5 symptom questions on 7-point scale ranging from 0 (no impairment) to 6 (maximum impairment). Total score: mean of scores of all 7 questions; ranging from 0 (totally controlled) to 6 (severely uncontrolled), higher score indicated lower asthma control. LS means and SE were derived from MMRM model with change from baseline in ACQ-7-IA values up to Week 52 as response variable, and treatment, age, baseline weight group, region, baseline eosinophil level, baseline FeNO level, baseline ICS dose level, visit, treatment by-visit interaction, baseline ACQ-7-IA value and baseline-by-visit interaction as covariates.
Time Frame: Baseline, Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 110 | 227
score on a scale | -0.99 (0.07) | -1.32 (0.05)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab; [analysis description as in outcome 5, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.0001, Mixed-effect model with repeated measure — Threshold for statistical significance at 5% significant level; LS mean difference = -0.33, 95% CI 2-sided [-0.50 to -0.16]

7. Secondary Outcome: Change From Baseline in Fractional Exhaled Nitric Oxide Level at Week 12: Baseline Blood Eosinophils >=300 Cells Per Microliter Population
Description: FeNO is a surrogate marker for airway inflammation. FeNO was analyzed using a NIOX instrument or similar analyzer using a flow rate of 50 mL/second, and reported in ppb. LS means and SE were derived from MMRM model with change from baseline in FeNO up to Week 12 as the response variable, and treatment, age, baseline weight group, region, baseline eosinophil level, baseline ICS level, visit, treatment by-visit interaction, baseline FeNO value and baseline-by-visit interaction as covariates.
Time Frame: Baseline, Week 12
Population: Analysis was performed on baseline blood eosinophils >=300 cells per microliter population. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: parts per billion
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 80 | 165
parts per billion | -0.81 (1.69) | -21.40 (1.21)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab; P-value and LS mean difference were derived from MMRM model with change from baseline in FeNO up to Week 12 as the response variable, and treatment, age, weight group, region, baseline eosinophil level, baseline ICS dose level, visit, treatment by-visit interaction, baseline FeNO value and baseline-by-visit interaction as covariates; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.0001, Mixed-effect model with repeated measure — Threshold for statistical significance at 5% significant level; LS mean difference = -20.59, 95% CI 2-sided [-24.60 to -16.59]

8. Secondary Outcome: Change From Baseline in Fractional Exhaled Nitric Oxide Level at Week 12: Type 2 Inflammatory Asthma Phenotype Population
Description: as for outcome 7
Time Frame: Baseline, Week 12
Population: Analysis was performed on type 2 inflammatory asthma phenotype population. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: parts per billion
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 110 | 226
parts per billion | -1.13 (1.43) | -18.97 (1.04)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab; [analysis description as in outcome 7, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.0001, Mixed-effect model with repeated measure — Threshold for statistical significance at 5% significant level; LS mean difference = -17.84, 95% CI 2-sided [-21.05 to -14.63]

9. Secondary Outcome: Change From Baseline in Pre-bronchodilator Percent Predicted Forced Expiratory Volume in 1 Second at Weeks 2, 4, 8, 24, 36 and 52: Type 2 Inflammatory Asthma Phenotype Population
Description: FEV1 was the volume of air (in liters) exhaled from the lungs in the first second of a forced expiration as measured by spirometer. LS means and SE were derived from MMRM model with change from baseline in pre-bronchodilator % predicted FEV1 values up to Week 52 as the response variable, and treatment, baseline weight group, region, ethnicity, baseline eosinophil level, baseline FeNO level, baseline ICS dose level, visit, treatment by-visit interaction, baseline % predicted FEV1 value and baseline-by-visit interaction as covariates.
Time Frame: Baseline, Weeks 2, 4, 8, 24, 36, 52
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: percent predicted FEV1
Groups:
- Placebo: Placebo (for Dupilumab), SC injection q2w for 52 weeks in combination with stable-dose background therapy of medium-dose ICS with a second controller medication (i.e., LABA, LAMA, LTRA or methylxanthines) or high-dose ICS alone or high-dose ICS with second controller. Albuterol/salbutamol or levalbuterol/levosalbutamol was given as reliever medication. Participants were followed up for 12 weeks after last dose (i.e. up to Week 64).
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 110 | 229
percent predicted FEV1
  Change at Week 2 | 4.84 (1.29) | 8.11 (0.95)
  Change at Week 4 | 3.55 (1.30) | 9.97 (0.97)
  Change at Week 8 | 4.27 (1.29) | 10.27 (0.96)
  Change at Week 24 | 4.27 (1.40) | 10.92 (1.04)
  Change at Week 36 | 6.63 (1.49) | 11.46 (1.10)
  Change at Week 52 | 4.36 (1.50) | 12.15 (1.10)

10. Secondary Outcome: Change From Baseline in Pre-bronchodilator Percent Predicted Forced Expiratory Volume in 1 Second at Weeks 2, 4, 8, 24, 36 and 52: Baseline Blood Eosinophils >=300 Cells Per Microliter Population
Description: as for outcome 9
Time Frame: Baseline, Weeks 2, 4, 8, 24, 36, 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: percent predicted of FEV1
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 80 | 168
percent predicted of FEV1
  Change at Week 2 | 3.94 (1.51) | 7.49 (1.08)
  Change at Week 4 | 2.19 (1.53) | 9.09 (1.12)
  Change at Week 8 | 2.48 (1.42) | 9.75 (1.04)
  Change at Week 24 | 3.45 (1.63) | 11.10 (1.19)
  Change at Week 36 | 6.87 (1.81) | 11.47 (1.31)
  Change at Week 52 | 4.08 (1.80) | 12.43 (1.30)

11. Secondary Outcome: Time to First Severe Exacerbation Event: Kaplan-Meier Estimates During 52-week Treatment Period: Type 2 Inflammatory Asthma Phenotype Population
Description: The time to first severe exacerbation was defined as date of the first severe exacerbation event - randomization date +1. A severe asthma exacerbation event was defined as a deterioration of asthma during the 52-week treatment period requiring: use of systemic corticosteroids for >=3 days; and/or hospitalization related to asthma symptoms or emergency room visit because of asthma requiring systemic corticosteroid treatment. Kaplan-Meier method was used for analysis.
Time Frame: Baseline up to Week 52
Population: Analysis was performed on type 2 inflammatory asthma phenotype population.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 114 | 236
days | NA [366.00 to NA] — Median and upper limit of 95% confidence interval (CI) was not estimable due to less than 50% of participants with events. | NA [NA to NA] — Median, lower and upper limit of 95 % CI was not estimable due to less than 50% of participants with events.

12. Secondary Outcome: Time to First Severe Exacerbation Event: Kaplan-Meier Estimates During 52-week Treatment Period: Baseline Blood Eosinophils >=300 Cells Per Microliter Population
Description: as for outcome 11
Time Frame: Baseline up to Week 52
Population: Analysis was performed on baseline blood eosinophils >=300 cells per microliter population.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 84 | 175
days | 366.0 [265.00 to NA] — Upper limit of 95 % CI was not estimable due to less than 50% of participants with events. | NA [NA to NA] — Median, lower and upper limit of 95 % CI was not estimable due to less than 50% of participants with events.

13. Secondary Outcome: Time to First Loss of Asthma Control (LOAC) Event: Kaplan-Meier Estimates During 52-week Treatment Period: Type 2 Inflammatory Asthma Phenotype Population
Description: Time to first LOAC event was date of first LOAC event - first dose date +1. A LOAC event was defined as deterioration of asthma during 52-week treatment period that resulted in any of the following: >= 6 additional reliever puffs of salbutamol/albuterol or levosalbutamol/levalbuterol in 24-hour period (compared to baseline) on 2 consecutive days; increase in ICS dose >=4 times than dose at Visit 2 (Week 0); a decrease in ante meridiem (AM)/post meridiem (PM) peak flow of 30% or more on 2 consecutive days of treatment, based on defined stability limit (defined as respective mean AM/PM peak expiratory flow obtained over last 7 days prior to randomization (Day 1); severe exacerbation event. Kaplan-Meier method was used for analysis.
Time Frame: Baseline up to Week 52
Population: Analysis was performed on type 2 inflammatory asthma phenotype population.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 114 | 236
days | 63.5 [42.00 to 84.00] | 140.0 [103.00 to 217.00]

14. Secondary Outcome: Time to First Loss of Asthma Control Event: Kaplan-Meier Estimates During 52-week Treatment Period: Baseline Blood Eosinophils >=300 Cells Per Microliter Population
Description: Time to first LOAC event was date of first LOAC event - first dose date +1. A LOAC event was defined as deterioration of asthma during 52-week treatment period that resulted in any of the following: >= 6 additional reliever puffs of salbutamol/albuterol or levosalbutamol/levalbuterol in 24-hour period (compared to baseline) on 2 consecutive days; increase in ICS dose >=4 times than dose at Visit 2 (Week 0); a decrease in AM/PM peak flow of 30% or more on 2 consecutive days of treatment, based on defined stability limit (defined as respective mean AM/PM peak expiratory flow obtained over last 7 days prior to randomization (Day 1); severe exacerbation event. Kaplan-Meier method was used for analysis.
Time Frame: Baseline up to Week 52
Population: Analysis was performed on baseline blood eosinophils >=300 cells per microliter population.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 84 | 175
days | 47.5 [38.00 to 84.00] | 135.0 [82.00 to 219.00]

15. Secondary Outcome: Absolute Change From Baseline in Pre-Bronchodilator FEV1 at Weeks 2, 4, 8, 12, 24, 36, 52: Type 2 Inflammatory Asthma Phenotype Population
Description: FEV1 was the volume of air (in liters) exhaled from the lungs in the first second of a forced expiration as measured by spirometer. LS means and SE were derived from MMRM model with change from baseline in pre-bronchodilator FEV1 values up to Week 52 as the response variable, and treatment, age, baseline weight group, region, sex, ethnicity, baseline height, baseline eosinophil level, baseline FeNO level, baseline ICS dose level, visit, treatment by-visit interaction, baseline pre-bronchodilator FEV1 value and baseline-by-visit interaction as covariates.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 24, 36, 52
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 110 | 229
liters
  Change at Week 2 | 0.08 (0.03) | 0.14 (0.02)
  Change at Week 4 | 0.06 (0.03) | 0.18 (0.02)
  Change at Week 8 | 0.09 (0.03) | 0.21 (0.02)
  Change at Week 12 | 0.12 (0.03) | 0.22 (0.02)
  Change at Week 24 | 0.14 (0.03) | 0.27 (0.02)
  Change at Week 36 | 0.23 (0.03) | 0.33 (0.02)
  Change at Week 52 | 0.24 (0.03) | 0.41 (0.02)

16. Secondary Outcome: Absolute Change From Baseline in Pre-Bronchodilator FEV1 at Weeks 2, 4, 8, 12, 24, 36, 52: Baseline Blood Eosinophils >=300 Cells Per Microliter Population
Description: as for outcome 15
Time Frame: Baseline, Weeks 2, 4, 8, 12, 24, 36, 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 80 | 168
liters
  Change at Week 2 | 0.07 (0.03) | 0.13 (0.02)
  Change at Week 4 | 0.04 (0.03) | 0.17 (0.02)
  Change at Week 8 | 0.06 (0.03) | 0.20 (0.02)
  Change at Week 12 | 0.12 (0.03) | 0.22 (0.02)
  Change at Week 24 | 0.13 (0.03) | 0.28 (0.03)
  Change at Week 36 | 0.24 (0.04) | 0.33 (0.03)
  Change at Week 52 | 0.25 (0.04) | 0.42 (0.03)

17. Secondary Outcome: Percent Change From Baseline in Pre-Bronchodilator Percent Predicted FEV1 at Weeks 2, 4, 8, 12, 24, 36, 52: Type 2 Inflammatory Asthma Phenotype Population
Description: as for outcome 9
Time Frame: Baseline, Weeks 2, 4, 8, 12, 24, 36, 52
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 110 | 229
percent change
  Change at Week 2 | 8.07 (2.00) | 13.38 (1.47)
  Change at Week 4 | 6.73 (2.10) | 16.01 (1.55)
  Change at Week 8 | 7.68 (1.87) | 16.33 (1.41)
  Change at Week 12 | 8.87 (2.10) | 16.94 (1.56)
  Change at Week 24 | 7.66 (2.12) | 17.61 (1.57)
  Change at Week 36 | 10.88 (2.85) | 19.19 (2.06)
  Change at Week 52 | 7.92 (2.81) | 20.06 (2.03)

18. Secondary Outcome: Percent Change From Baseline in Pre-Bronchodilator Percent Predicted FEV1 at Weeks 2, 4, 8, 12, 24, 36, 52: Baseline Blood Eosinophils >=300 Cells Per Microliter Population
Description: as for outcome 9
Time Frame: Baseline, Weeks 2, 4, 8, 12, 24, 36, 52
Population: Analysis was performed on baseline blood eosinophils >=300 cells per microliter population . Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 80 | 168
percent change
  Change at Week 2 | 7.55 (2.41) | 12.76 (1.73)
  Change at Week 4 | 5.81 (2.57) | 15.20 (1.87)
  Change at Week 8 | 6.09 (2.10) | 16.01 (1.56)
  Change at Week 12 | 9.56 (2.45) | 17.14 (1.79)
  Change at Week 24 | 7.44 (2.54) | 18.09 (1.85)
  Change at Week 36 | 12.15 (3.67) | 19.65 (2.61)
  Change at Week 52 | 8.50 (3.58) | 20.97 (2.54)

19. Secondary Outcome: Change From Baseline in Morning (AM) Peak Expiratory Flow (PEF) at Weeks 2, 4, 8, 12, 24, 36, and 52: Type 2 Inflammatory Asthma Phenotype Population
Description: The PEF is a participant's maximum speed of expiration, as measured with a peak flow meter. Peak flow testing for AM PEF was performed in morning prior to taking any salbutamol/albuterol or levosalbutamol/levalbuterol reliever medication. Baseline AM PEF was the mean AM measurement recorded for the 7 days prior to the first dose of investigational product. LS means and SE were derived from MMRM model with change from baseline in AM PEF (liters/minute) values up to Week 52 as the response variable, and treatment, age, baseline weight group, region, baseline eosinophil level, baseline FeNO level, baseline ICS dose level, visit, treatment by-visit interaction, baseline AM PEF (liters/minute) value and baseline-by-visit interaction as covariates.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 24, 36, 52
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: liters/minute
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 110 | 228
liters/minute
  Change at Week 2 | 5.57 (2.66) | 6.50 (2.00)
  Change at Week 4 | 7.10 (3.31) | 12.81 (2.43)
  Change at Week 8 | 7.37 (3.56) | 18.05 (2.59)
  Change at Week 12 | 5.37 (3.93) | 19.38 (2.85)
  Change at Week 24 | 8.76 (4.53) | 23.32 (3.25)
  Change at Week 36 | 17.70 (4.99) | 26.77 (3.56)
  Change at Week 52 | 19.88 (5.16) | 31.45 (3.69)

20. Secondary Outcome: Change From Baseline in Evening (PM) Peak Expiratory Flow at Weeks 2, 4, 8, 12, 24, 36, and 52: Type 2 Inflammatory Asthma Phenotype Population
Description: The PEF is a participant's maximum speed of expiration, as measured with a peak flow meter. Peak flow testing for PM PEF was performed in evening prior to taking any salbutamol/albuterol or levosalbutamol/levalbuterol reliever medication. Baseline PM PEF was the mean PM measurement recorded for the 7 days prior to the first dose of investigational product. LS means and SE were derived from MMRM model with change from baseline in PM PEF (liters/minute) values up to Week 52 as the response variable, and treatment, age, baseline weight group, region, baseline eosinophil level, baseline FeNO level, baseline ICS dose level, visit, treatment by-visit interaction, baseline PM PEF (liters/minute) value and baseline-by-visit interaction as covariates.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 24, 36, 52
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: liters/minute
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 110 | 228
liters/minute
  Change at Week 2 | 7.62 (2.94) | 10.60 (2.20)
  Change at Week 4 | 6.92 (3.42) | 15.23 (2.52)
  Change at Week 8 | 5.52 (3.60) | 20.17 (2.64)
  Change at Week 12 | 1.71 (3.92) | 19.68 (2.85)
  Change at Week 24 | 3.78 (4.61) | 22.75 (3.32)
  Change at Week 36 | 12.55 (5.06) | 24.69 (3.62)
  Change at Week 52 | 16.46 (5.20) | 28.20 (3.73)

21. Secondary Outcome: Change From Baseline in Morning (AM) Peak Expiratory Flow at Weeks 2, 4, 8, 12, 24, 36, and 52: Baseline Blood Eosinophils >=300 Cells Per Microliter Population
Description: as for outcome 19
Time Frame: Baseline, Weeks 2, 4, 8, 12, 24, 36, 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: liters/minute
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 80 | 167
liters/minute
  Change at Week 2 | 5.85 (2.97) | 7.94 (2.21)
  Change at Week 4 | 5.62 (3.80) | 11.75 (2.76)
  Change at Week 8 | 5.54 (4.09) | 17.32 (2.96)
  Change at Week 12 | 4.77 (4.65) | 19.25 (3.34)
  Change at Week 24 | 4.78 (5.05) | 23.62 (3.61)
  Change at Week 36 | 14.80 (5.77) | 26.78 (4.08)
  Change at Week 52 | 19.75 (6.33) | 32.80 (4.49)

22. Secondary Outcome: Change From Baseline in Evening (PM) Peak Expiratory Flow at Weeks 2, 4, 8, 12, 24, 36, and 52: Baseline Blood Eosinophils >=300 Cells Per Microliter Population
Description: as for outcome 20
Time Frame: Baseline, Weeks 2, 4, 8, 12, 24, 36, 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: liters/minute
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 80 | 167
liters/minute
  Change at Week 2 | 5.64 (3.42) | 10.02 (2.53)
  Change at Week 4 | 4.36 (3.96) | 13.09 (2.89)
  Change at Week 8 | 0.92 (4.05) | 17.51 (2.96)
  Change at Week 12 | -1.37 (4.57) | 17.73 (3.30)
  Change at Week 24 | -1.37 (5.21) | 20.30 (3.74)
  Change at Week 36 | 7.52 (6.01) | 23.23 (4.26)
  Change at Week 52 | 14.67 (6.39) | 26.60 (4.54)

23. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC) at Weeks 2, 4, 8, 12, 24, 36, 52: Type 2 Inflammatory Asthma Phenotype Population
Description: FVC is a standard pulmonary function test used to quantify respiratory muscle weakness. FVC is the volume of air (in liters) that can be forcibly blown out after full inspiration in the upright position, measured in liters. LS means and SE were derived from MMRM model with change from baseline in FVC values up to Week 52 as the response variable, and treatment, age, baseline weight group, region, sex, ethnicity, baseline height, baseline eosinophil level, baseline FeNO level, baseline ICS dose level, visit, treatment by-visit interaction, baseline FVC value and baseline-by-visit interaction as covariates.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 24, 36, 52
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 110 | 229
liters
  Change at Week 2 | 0.07 (0.02) | 0.07 (0.02)
  Change at Week 4 | 0.07 (0.03) | 0.11 (0.02)
  Change at Week 8 | 0.10 (0.02) | 0.13 (0.02)
  Change at Week 12 | 0.12 (0.03) | 0.14 (0.02)
  Change at Week 24 | 0.16 (0.03) | 0.20 (0.02)
  Change at Week 36 | 0.22 (0.03) | 0.28 (0.02)
  Change at Week 52 | 0.27 (0.03) | 0.37 (0.02)

24. Secondary Outcome: Change From Baseline in Forced Vital Capacity at Weeks 2, 4, 8, 12, 24, 36, 52: Baseline Blood Eosinophils >=300 Cells Per Microliter Population
Description: as for outcome 23
Time Frame: Baseline, Weeks 2, 4, 8, 12, 24, 36, 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 80 | 168
liters
  Change at Week 2 | 0.07 (0.03) | 0.06 (0.02)
  Change at Week 4 | 0.08 (0.03) | 0.09 (0.02)
  Change at Week 8 | 0.09 (0.03) | 0.13 (0.02)
  Change at Week 12 | 0.13 (0.03) | 0.14 (0.02)
  Change at Week 24 | 0.17 (0.03) | 0.22 (0.03)
  Change at Week 36 | 0.24 (0.04) | 0.28 (0.03)
  Change at Week 52 | 0.29 (0.04) | 0.38 (0.03)

25. Secondary Outcome: Change From Baseline in Forced Expiratory Flow (FEF) 25-75% at Weeks 2, 4, 8, 12, 24, 36, 52: Type 2 Inflammatory Asthma Phenotype Population
Description: FEF is the amount of air (in liters) which can be forcibly exhaled from the lungs in the first second of a forced exhalation. FEF 25-75% was defined as the mean FEF between 25% and 75% of the FVC, where FVC was defined as the volume of air (in liters) that can be forcibly blown out after full inspiration in the upright position. LS means and SE were derived from MMRM model with change from baseline in FEF 25-75% values up to Week 52 as the response variable, and treatment, age, baseline weight group, region, sex, ethnicity, baseline height, baseline eosinophil level, baseline FeNO level, baseline ICS dose level, visit, treatment by-visit interaction, baseline FEF 25-75% value and baseline-by-visit interaction as covariates.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 24, 36, 52
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: liters/second
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 110 | 229
liters/second
  Change at Week 2 | 0.11 (0.05) | 0.28 (0.04)
  Change at Week 4 | 0.07 (0.05) | 0.34 (0.04)
  Change at Week 8 | 0.10 (0.05) | 0.39 (0.04)
  Change at Week 12 | 0.14 (0.05) | 0.41 (0.04)
  Change at Week 24 | 0.16 (0.05) | 0.44 (0.04)
  Change at Week 36 | 0.29 (0.05) | 0.49 (0.04)
  Change at Week 52 | 0.29 (0.06) | 0.60 (0.04)

26. Secondary Outcome: Change From Baseline in Forced Expiratory Flow 25-75% at Weeks 2, 4, 8, 12, 24, 36, 52: Baseline Blood Eosinophils >=300 Cells Per Microliter Population
Description: FEF is the amount of air (in liters) which can be forcibly exhaled from the lungs in the first second of a forced exhalation. FEF 25-75% was defined as the mean FEF between 25% and 75% of the FVC, where FVC was defined as the volume of air (in liters) that can be forcibly blown out after full inspiration in the upright position. LS means and SE were derived from MMRM model with change from baseline in FE F25-75% values up to Week 52 as the response variable, and treatment, age, baseline weight group, region, sex, ethnicity, baseline height, baseline eosinophil level, baseline FeNO level, baseline ICS dose level, visit, treatment by-visit interaction, baseline FEF 25-75% value and baseline-by-visit interaction as covariates.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 24, 36, 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: liters/second
Groups:
- Placebo: Placebo (for Dupilumab), SC injection q2w for 52 weeks in combination with stable-dose background therapy of medium-dose ICS with a second controller medication (i.e., LABA, LAMA, LTRA or methylxanthines) or high-dose ICS alone or high-dos medication ICS with second controller. Albuterol/salbutamol or levalbuterol/levosalbutamol was given as reliever medication. Participants were followed up for 12 weeks after last dose (i.e. up to Week 64).
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 80 | 168
liters/second
  Change at Week 2 | 0.07 (0.05) | 0.29 (0.04)
  Change at Week 4 | 0.00 (0.05) | 0.33 (0.04)
  Change at Week 8 | 0.02 (0.06) | 0.40 (0.04)
  Change at Week 12 | 0.10 (0.05) | 0.42 (0.04)
  Change at Week 24 | 0.12 (0.06) | 0.47 (0.04)
  Change at Week 36 | 0.27 (0.06) | 0.51 (0.05)
  Change at Week 52 | 0.26 (0.07) | 0.65 (0.05)

27. Secondary Outcome: Change From Baseline in Post-Bronchodilator FEV1 at Weeks 2, 4, 8, 12, 24, 36, and 52: Type 2 Inflammatory Asthma Phenotype Population
Description: Participants were assessed for post-bronchodilator FEV1 30 minutes after bronchodilator administration (200 to 400 mg [2 to 4 puffs] of albuterol/salbutamol or 45 to 90 micrograms [2 to 4 puffs] of levalbuterol/levosalbutamol). FEV1 was the volume of air (in liters) exhaled in the first second of a forced expiration as measured by spirometer. LS means and SE were derived from MMRM model with change from baseline in post-bronchodilator FEV1 values up to Week 52 as the response variable, and treatment, baseline weight group, region, ethnicity, baseline eosinophil level, baseline FeNO level, baseline ICS dose level, visit, treatment by-visit interaction, baseline post-bronchodilator FEV1 value and baseline-by-visit interaction as covariates.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 24, 36, 52
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 110 | 230
liters
  Change at Week 2 | 0.61 (1.26) | 1.51 (0.92)
  Change at Week 4 | -0.02 (1.15) | 2.42 (0.86)
  Change at Week 8 | -0.79 (1.21) | 2.85 (0.90)
  Change at Week 12 | -0.32 (1.23) | 2.48 (0.91)
  Change at Week 24 | -0.50 (1.31) | 2.60 (0.96)
  Change at Week 36 | 0.55 (1.46) | 3.15 (1.07)
  Change at Week 52 | -0.75 (1.48) | 3.62 (1.08)

28. Secondary Outcome: Change From Baseline in Post-Bronchodilator FEV1 at Weeks 2, 4, 8, 12, 24, 36, and 52: Baseline Blood Eosinophils >=300 Cells Per Microliter Population
Description: as for outcome 27
Time Frame: Baseline, Weeks 2, 4, 8, 12, 24, 36, 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 80 | 169
liters
  Change at Week 2 | 0.10 (1.49) | 0.52 (1.07)
  Change at Week 4 | -0.29 (1.35) | 1.44 (1.00)
  Change at Week 8 | -2.05 (1.31) | 1.81 (0.98)
  Change at Week 12 | -0.61 (1.44) | 2.28 (1.04)
  Change at Week 24 | -0.80 (1.54) | 2.25 (1.12)
  Change at Week 36 | 0.72 (1.80) | 2.87 (1.31)
  Change at Week 52 | -0.52 (1.79) | 3.13 (1.30)

29. Secondary Outcome: Change From Baseline in Morning Asthma Symptom Score at Weeks 2, 4, 8, 12, 24, 36, and 52: Type 2 Inflammatory Asthma Phenotype Population
Description: The morning asthma symptom score evaluated participant's overall asthma symptoms experienced during the previous night. It ranged from 0 (no asthma symptoms, slept through the night) to 4 (bad night, awake most of the night because of asthma), where lower scores indicate more mild symptoms and higher scores indicate more severe symptoms. LS means and SE were derived from MMRM model with change from baseline in AM asthma symptom score values up to Week 52 as the response variable, and treatment, age, baseline weight group, region, baseline eosinophil level, baseline FeNO level, baseline ICS dose level, visit, treatment by-visit interaction, baseline AM asthma symptom score value and baseline-by-visit interaction as covariates.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 24, 36, 52
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 110 | 228
score on a scale
  Change at Week 2 | -0.22 (0.04) | -0.18 (0.03)
  Change at Week 4 | -0.29 (0.05) | -0.34 (0.04)
  Change at Week 8 | -0.37 (0.05) | -0.39 (0.04)
  Change at Week 12 | -0.34 (0.05) | -0.48 (0.04)
  Change at Week 24 | -0.46 (0.05) | -0.56 (0.04)
  Change at Week 36 | -0.48 (0.05) | -0.56 (0.04)
  Change at Week 52 | -0.50 (0.05) | -0.61 (0.04)

30. Secondary Outcome: Change From Baseline in Evening Asthma Symptom Score at Weeks 2, 4, 8, 12, 24, 36, and 52: Type 2 Inflammatory Asthma Phenotype Population
Description: The evening asthma symptom score evaluated participant's overall asthma symptoms experienced during the day. It ranged from 0 (very well, no asthma symptoms) to 4 (asthma very bad, unable to carry out daily activities as usual), where lower scores indicate more mild symptoms and higher scores indicate more severe symptoms. LS means and SE were derived from MMRM model with change from baseline in PM asthma symptom score values up to Week 52 as response variable, and treatment, age, baseline weight group, region, baseline eosinophil level, baseline FeNO level, baseline ICS dose level, visit, treatment by-visit interaction, baseline PM asthma symptom score value and baseline-by-visit interaction as covariates.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 24, 36, 52
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 110 | 228
score on a scale
  Change at Week 2 | -0.17 (0.05) | -0.13 (0.03)
  Change at Week 4 | -0.25 (0.05) | -0.29 (0.04)
  Change at Week 8 | -0.33 (0.06) | -0.40 (0.04)
  Change at Week 12 | -0.30 (0.06) | -0.45 (0.04)
  Change at Week 24 | -0.44 (0.06) | -0.53 (0.04)
  Change at Week 36 | -0.47 (0.06) | -0.55 (0.04)
  Change at Week 52 | -0.50 (0.06) | -0.59 (0.04)

31. Secondary Outcome: Change From Baseline in Morning Asthma Symptom Score at Weeks 2, 4, 8, 12, 24, 36, and 52: Baseline Blood Eosinophils >=300 Cells Per Microliter Population
Description: as for outcome 29
Time Frame: Baseline, Weeks 2, 4, 8, 12, 24, 36, 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 80 | 167
score on a scale
  Change at Week 2 | -0.24 (0.05) | -0.20 (0.04)
  Change at Week 4 | -0.32 (0.06) | -0.34 (0.04)
  Change at Week 8 | -0.38 (0.06) | -0.40 (0.05)
  Change at Week 12 | -0.33 (0.06) | -0.48 (0.04)
  Change at Week 24 | -0.45 (0.06) | -0.55 (0.04)
  Change at Week 36 | -0.46 (0.06) | -0.56 (0.04)
  Change at Week 52 | -0.50 (0.06) | -0.62 (0.04)

32. Secondary Outcome: Change From Baseline in Evening Asthma Symptom Score at Weeks 2, 4, 8, 12, 24, 36, and 52: Baseline Blood Eosinophils >=300 Cells Per Microliter Population
Description: as for outcome 30
Time Frame: Baseline, Weeks 2, 4, 8, 12, 24, 36, 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 80 | 167
score on a scale
  Change at Week 2 | -0.18 (0.05) | -0.15 (0.04)
  Change at Week 4 | -0.27 (0.06) | -0.29 (0.04)
  Change at Week 8 | -0.30 (0.06) | -0.41 (0.05)
  Change at Week 12 | -0.29 (0.07) | -0.48 (0.05)
  Change at Week 24 | -0.42 (0.06) | -0.53 (0.05)
  Change at Week 36 | -0.43 (0.06) | -0.56 (0.05)
  Change at Week 52 | -0.51 (0.06) | -0.60 (0.04)

33. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire-Interviewer Administered, 5-question Version (ACQ-5-IA) at Weeks 2, 4, 8, 12, 24, 36, and 52: Type 2 Inflammatory Asthma Phenotype Population
Description: ACQ-5-IA has 5 questions, reflecting top-scoring 5 asthma symptoms: frequency of nocturnal awakenings, severity of asthma symptoms in the mornings, limitation of daily activities, shortness of breath due to asthma and wheeze. Participants were asked to recall how their asthma had been during the previous week and to respond to each of the five symptom questions on a 7-point scale ranging from 0 (no impairment) to 6 (maximum impairment). ACQ-5-IA total score was mean of the scores of all 5 questions and, therefore, ranged from 0 (totally controlled) to 6 (severely uncontrolled), higher scores indicated lower asthma control. LS means and SE were derived from MMRM model with change from baseline in ACQ-5-IA values up to Week 52 as the response variable, and treatment, age, baseline weight group, region, baseline eosinophil level, baseline FeNO level, baseline ICS dose level, visit, treatment by-visit interaction, baseline ACQ-5-IA value and baseline-by-visit interaction as covariates.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 24, 36, 52
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 110 | 227
score on a scale
  Change at Week 2 | -0.72 (0.09) | -0.77 (0.06)
  Change at Week 4 | -0.86 (0.08) | -1.09 (0.06)
  Change at Week 8 | -1.04 (0.09) | -1.24 (0.07)
  Change at Week 12 | -1.04 (0.08) | -1.35 (0.06)
  Change at Week 24 | -1.18 (0.08) | -1.46 (0.06)
  Change at Week 36 | -1.25 (0.08) | -1.57 (0.06)
  Change at Week 52 | -1.30 (0.07) | -1.70 (0.05)

34. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire-Interviewer Administered, 5-question Version at Weeks 2, 4, 8, 12, 24, 36, and 52: Baseline Blood Eosinophils >=300 Cells Per Microliter Population
Description: as for outcome 33
Time Frame: Baseline, Weeks 2, 4, 8, 12, 24, 36, 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 80 | 166
score on a scale
  Change at Week 2 | -0.63 (0.11) | -0.76 (0.08)
  Change at Week 4 | -0.75 (0.10) | -1.10 (0.07)
  Change at Week 8 | -0.98 (0.10) | -1.27 (0.07)
  Change at Week 12 | -1.00 (0.10) | -1.37 (0.07)
  Change at Week 24 | -1.06 (0.09) | -1.48 (0.07)
  Change at Week 36 | -1.17 (0.09) | -1.59 (0.07)
  Change at Week 52 | -1.25 (0.08) | -1.71 (0.06)

35. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire-Interviewer Administered, 7-question Version at Weeks 2, 4, 8, 12, 36, and 52: Baseline Blood Eosinophils >=300 Cells Per Microliter Population
Description: ACQ-7-IA had 7 questions, assessed: frequency of nocturnal awakenings, severity of asthma symptoms in the mornings, limitation of daily activities, shortness of breath due to asthma and wheeze, reliever medication use, and FEV1 (% predicted). Participants recalled their previous week asthma and answered 5 symptom questions on 7-point scale ranging from 0 (no impairment) to 6 (maximum impairment). Total score:mean of scores of all 7 questions; ranging from 0 (totally controlled) to 6 (severely uncontrolled), higher score indicated lower asthma control. LS means and SE were derived from MMRM model with change from baseline in ACQ-7-IA values up to Week 52 as response variable and treatment, age, baseline weight group, region, baseline eosinophil level, baseline FeNO level, baseline ICS dose level, visit, treatment by-visit interaction, baseline ACQ-7-IA value and baseline-by-visit interaction as covariates.
Time Frame: Baseline, Weeks 2, 4, 8,12, 36, 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 80 | 166
score on a scale
  Change at Week 2 | -0.50 (0.09) | -0.70 (0.07)
  Change at Week 4 | -0.64 (0.09) | -1.02 (0.06)
  Change at Week 8 | -0.83 (0.09) | -1.16 (0.06)
  Change at Week 12 | -0.85 (0.09) | -1.24 (0.06)
  Change at Week 36 | -1.01 (0.08) | -1.43 (0.06)
  Change at Week 52 | -1.04 (0.08) | -1.54 (0.06)

36. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire-Interviewer Administered, 7-question Version at Weeks 2, 4, 8, 12, 36, and 52: Type 2 Inflammatory Asthma Phenotype Population
Description: ACQ-7-IA had 7 questions, assessed: frequency of nocturnal awakenings, severity of asthma symptoms in the mornings, limitation of daily activities due to asthma, shortness of breath due to asthma and wheeze, reliever medication use, and FEV1 (% predicted). Participants recalled their previous week asthma and answered 5 symptom questions on 7-point scale ranging from 0 (no impairment) to 6 (maximum impairment). Total score: mean of scores of all 7 questions; ranging from 0 (totally controlled) to 6 (severely uncontrolled), higher score indicated lower asthma control. LS means and SE were derived from MMRM model with change from baseline in ACQ-7-IA values up to Week 52 as response variable, and treatment, age, baseline weight group, region, baseline eosinophil level, baseline FeNO level, baseline ICS dose level, visit, treatment by-visit interaction, baseline ACQ-7-IA value and baseline-by-visit interaction as covariates.
Time Frame: Baseline, Weeks 2, 4, 8,12, 36, 52
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 110 | 227
score on a scale
  Change at Week 2 | -0.60 (0.08) | -0.72 (0.06)
  Change at Week 4 | -0.74 (0.07) | -1.03 (0.05)
  Change at Week 8 | -0.91 (0.08) | -1.14 (0.06)
  Change at Week 12 | -0.89 (0.07) | -1.23 (0.05)
  Change at Week 36 | -1.09 (0.07) | -1.41 (0.05)
  Change at Week 52 | -1.09 (0.06) | -1.53 (0.05)

37. Secondary Outcome: Change From Baseline in Number of Puffs of Reliever Medication Used Per 24 Hours at Weeks 2, 4, 8, 12, 24, 36, and 52: Type 2 Inflammatory Asthma Phenotype Population
Description: Participants might be administered salbutamol/albuterol or levosalbutamol/levalbuterol as reliever medication as needed. Number of reliever medication inhalations were recorded daily in electronic diary/PEF meter. When Nebulizer solutions were used as alternative delivery method, nebulizer dose was converted to number of puffs as per conversion factor: salbutamol/albuterol nebulizer solution (2.5 mg) and levosalbutamol/levalbuterol (1.25 mg) corresponds to 4 puffs. Change From Baseline in number of puffs of reliever medication used per 24 hours at specified weeks was reported. LS means and SE were derived from MMRM model with change from baseline in number of puffs of reliever medication/24 hours values up to Week 52 as response variable and treatment, age, baseline: weight group, region, eosinophil level, FeNO level, ICS dose level, visit, treatment by-visit interaction, baseline number of puffs of reliever medication/24 hours value and baseline-by-visit interaction as covariates.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 24, 36, 52
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: puffs of reliever medication per 24 hour
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 110 | 228
puffs of reliever medication per 24 hour
  Change at Week 2 | -0.78 (0.17) | -0.65 (0.12)
  Change at Week 4 | -0.99 (0.17) | -1.02 (0.13)
  Change at Week 8 | -1.24 (0.17) | -1.28 (0.13)
  Change at Week 12 | -0.93 (0.18) | -1.41 (0.13)
  Change at Week 24 | -1.43 (0.17) | -1.61 (0.13)
  Change at Week 36 | -1.37 (0.17) | -1.60 (0.13)
  Change at Week 52 | -1.59 (0.16) | -1.72 (0.12)

38. Secondary Outcome: Change From Baseline in Number of Puffs of Reliever Medication Used Per 24 Hours at Weeks 2, 4, 8, 12, 24, 36, and 52: Baseline Blood Eosinophils >=300 Cells Per Microliter Population
Description: as for outcome 37
Time Frame: Baseline, Weeks 2, 4, 8, 12, 24, 36, 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: puffs of reliever medication per 24 hour
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 80 | 167
puffs of reliever medication per 24 hour
  Change at Week 2 | -0.75 (0.19) | -0.67 (0.14)
  Change at Week 4 | -1.02 (0.20) | -1.01 (0.15)
  Change at Week 8 | -1.15 (0.20) | -1.29 (0.14)
  Change at Week 12 | -1.02 (0.20) | -1.39 (0.14)
  Change at Week 24 | -1.25 (0.20) | -1.53 (0.15)
  Change at Week 36 | -1.20 (0.21) | -1.49 (0.15)
  Change at Week 52 | -1.45 (0.19) | -1.58 (0.14)

39. Secondary Outcome: Change From Baseline in Number of Nocturnal Awakenings Per Night at Weeks 2, 4, 8, 12, 24, 36, and 52: Type 2 Inflammatory Asthma Phenotype Population
Description: Participants recorded every morning the number of asthma-related nocturnal awakenings requiring use of rescue medication that occurred during the previous night. Change from baseline in number of nocturnal awakenings per night at specified weeks was reported. LS means and SE were derived from MMRM model with change from baseline in number of nocturnal awakenings values up to Week 52 as the response variable, and treatment, age, baseline weight group, region, baseline eosinophil level, baseline FeNO level, baseline ICS dose level, visit, treatment by-visit interaction, baseline number of nocturnal awakenings value and baseline-by-visit interaction as covariates.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 24, 36, 52
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: nocturnal awakenings per night
Groups:
- Dupilumab: Dupilumab 200 mg (1.14 mL; for >30 kg bodyweight) or 100 mg (0.67 mL; for <=30 kg body weight), SC injection q2w for 50 weeks in combination with stable-dose background therapy of medium-dose ICS therapy with a second controller medication (i.e., LABA, LAMA, LTRA or methylxanthines) or high-dose ICS alone or high-dose ICS with second controller. Albuterol/salbutamol or levalbuterol/levosalbutamol was given as reliever medication. Participants were followed up for 12 weeks after last dose (i.e. up to Week 64).
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 110 | 228
nocturnal awakenings per night
  Change at Week 2 | -0.13 (0.03) | -0.13 (0.02)
  Change at Week 4 | -0.16 (0.03) | -0.21 (0.03)
  Change at Week 8 | -0.21 (0.04) | -0.21 (0.03)
  Change at Week 12 | -0.17 (0.04) | -0.26 (0.03)
  Change at Week 24 | -0.23 (0.03) | -0.29 (0.02)
  Change at Week 36 | -0.25 (0.03) | -0.29 (0.02)
  Change at Week 52 | -0.26 (0.03) | -0.32 (0.02)

40. Secondary Outcome: Change From Baseline in Number of Nocturnal Awakenings Per Night at Weeks 2, 4, 8, 12, 24, 36, and 52: Baseline Blood Eosinophils >=300 Cells Per Microliter Population
Description: as for outcome 39
Time Frame: Baseline, Weeks 2, 4, 8, 12, 24, 36, 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: nocturnal awakenings per night
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 80 | 167
nocturnal awakenings per night
  Change at Week 2 | -0.15 (0.03) | -0.12 (0.02)
  Change at Week 4 | -0.19 (0.04) | -0.21 (0.03)
  Change at Week 8 | -0.22 (0.05) | -0.20 (0.04)
  Change at Week 12 | -0.16 (0.04) | -0.25 (0.03)
  Change at Week 24 | -0.21 (0.04) | -0.28 (0.03)
  Change at Week 36 | -0.25 (0.04) | -0.27 (0.03)
  Change at Week 52 | -0.26 (0.03) | -0.32 (0.02)

41. Secondary Outcome: Change From Baseline in Pediatric Asthma Quality of Life (QoL) Questionnaire With Standardized Activities-Interviewer Administered (PAQLQ[S] IA) Scores at Weeks 12, 24, 36, and 52: Type 2 Inflammatory Asthma Phenotype Population
Description: PAQLQ(S)-IA, a disease-specific, interviewer-administered QoL questionnaire designed to measure functional impairments that are most important to children >=7 years with asthma. The PAQLQ(S)-IA comprises of 23 items in 3 domains: symptoms (10 items), activity limitation (5 items) and emotional function (8 items). Each item was scored on a 7-point likert scale (1=maximal impairment to 7=no impairment). 23 items of questionnaire were averaged to produce 1 overall quality of life score ranging from 1 (severely impaired) to 7 (not impaired at all), higher scores indicated better quality of life. LS means and SE were derived from MMRM model with change from baseline in PAQLQ(S)-IA global score values up to Week 52 as the response variable, and treatment, age, baseline weight group, region, baseline eosinophil level, baseline FeNO level, baseline ICS dose level, visit, treatment by-visit interaction, baseline PAQLQ(S)-IA global score value and baseline-by-visit interaction as covariates.
Time Frame: Baseline, Weeks 12, 24, 36, 52
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 102 | 201
score on a scale
  Change at Week 12 | 0.97 (0.09) | 1.08 (0.07)
  Change at Week 24 | 1.11 (0.09) | 1.30 (0.07)
  Change at Week 36 | 1.15 (0.09) | 1.48 (0.07)
  Change at Week 52 | 1.19 (0.08) | 1.53 (0.06)

42. Secondary Outcome: Change From Baseline in Pediatric Asthma Quality of Life Questionnaire With Standardized Activities-Interviewer Administered Scores at Weeks 12, 24, 36, and 52: Baseline Blood Eosinophils >=300 Cells Per Microliter Population
Description: as for outcome 41
Time Frame: Baseline, Weeks 12, 24, 36, 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 76 | 149
score on a scale
  Change at Week 12 | 0.90 (0.10) | 1.11 (0.08)
  Change at Week 24 | 1.06 (0.10) | 1.36 (0.08)
  Change at Week 36 | 1.07 (0.10) | 1.51 (0.08)
  Change at Week 52 | 1.23 (0.09) | 1.56 (0.07)

43. Secondary Outcome: Healthcare Resource Utilization (HCRU): Number of School and Work Days Missed Due to LOAC: Type 2 Inflammatory Asthma Phenotype Population
Description: The number of days missed from school by the participant and the number of days missed from work by the caregiver of participant due to a LOAC were collected in the electronic-case report form (eCRF). Cumulative number of missed days (school days and work days) up to week 52 were computed and summarized using mean and standard deviation (SD).
Time Frame: Baseline to Week 52
Population: Analysis was performed on type 2 inflammatory asthma phenotype population. For the caregiver data, population assessed was children participant only and the work days missed by their caregiver were counted.
Measure: Mean (Standard Deviation); unit: days
Groups:
- Placebo: Placebo (for Dupilumab), SC injection q2w for 50 weeks in combination with stable-dose background therapy of medium-dose ICS therapy with a second controller medication (i.e., LABA, LAMA, LTRA or methylxanthines) or high-dose ICS alone or high-dose ICS with second controller medication. Albuterol/salbutamol or levalbuterol/levosalbutamol was given as reliever medication. Participants were followed up for 12 weeks after last dose (i.e. up to Week 64).
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 114 | 236
days
  Number of missed school days | 2.1 (4.2) | 1.0 (2.3)
  Number of missed work days | 0.7 (1.9) | 0.2 (0.8)

44. Secondary Outcome: Healthcare Resource Utilization: Number of School and Work Days Missed Due to LOAC: Baseline Blood Eosinophils >=300 Cells Per Microliter Population
Description: The number of days missed from school by the participant and the number of days missed from work by the caregiver of participant due to a LOAC were collected in the eCRF. Cumulative number of missed days (school days and work days) up to week 52 were computed and summarized using mean and SD.
Time Frame: Baseline to Week 52
Population: Analysis was performed on baseline blood eosinophils >=300 cells per microliter population. For the caregiver data, population assessed was children participant only and the work days missed by their caregiver were counted.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 84 | 175
days
  Number of missed school days | 2.0 (3.5) | 0.9 (2.0)
  Number of missed work days | 0.6 (1.8) | 0.2 (0.7)

45. Secondary Outcome: Healthcare Resource Utilization: Percentage of Participants Who Had Missed Greater Than or Equal to 5 School/Work Days Due to LOAC: Type 2 Inflammatory Asthma Phenotype Population
Description: The number of days missed from school for the participant and the missed number of days from work for the caregiver due to a LOAC were collected in the eCRF. The percentage of participants who had at least 5 days (school days and work days) missed due to LOAC over the study period was reported.
Time Frame: Baseline to Week 52
Population: as for outcome 43
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 114 | 236
percentage of participants
  Percentage of participants with >=5 missed school days | 17.5 | 9.7
  Percentage of participants with >=5 missed work days | 7 | 0.8

46. Secondary Outcome: Healthcare Resource Utilization: Percentage of Participants Who Had Missed Greater Than or Equal to 5 School/Work Days Due to LOAC: Baseline Blood Eosinophils >=300 Cells Per Microliter Population
Description: as for outcome 45
Time Frame: Baseline to Week 52
Population: as for outcome 44
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 84 | 175
percentage of participants
  Percentage of participants with >=5 missed school days | 17.9 | 8.6
  Percentage of participants with >=5 missed work days | 6 | 0.6

47. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: Adverse event (AE) was defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and did not necessary have to had a causal relationship with treatment.TEAEs were defined as AEs that developed or worsened in grade or became serious during TEAE period which was defined as the period from the time of first dose of study drug to the end of post-treatment period. A serious adverse events (SAE) was any untoward medical occurrence that at any dose resulted in: death; or life-threatening experience; or required inpatient hospitalization or prolongation of existing hospitalization; or resulted in persistent or significant disability/incapacity; or was a congenital anomaly/birth defect or a medically important event. TEAEs included both SAEs and non-SAEs.
Time Frame: From Baseline up to Week 64
Population: Analysis was performed on safety population which included all participants who actually received at least 1 dose or part of a dose of IMP and were analyzed according to the actually treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 134 | 271
Participants
  Any TEAE | 107 | 225
  TESAE | 6 | 13

48. Secondary Outcome: Pharmacokinetics (PK) Assessment: Functional Dupilumab Concentration in Serum
Description: Data for this outcome measure was planned to be collected and analyzed separately for dupilumab 100 mg and 200 mg dose and not planned to be collected and analyzed for placebo arm.
Time Frame: Baseline, Weeks 6, 12, 24, 52, 64
Population: Analysis was performed on the PK population which consisted of all participants who actually received at least 1 dose or part of a dose of the IMP, analyzed according to the treatment actually received with at least one non-missing result for functional dupilumab concentration in serum. Here, 'number analyzed'=number of participants with available data for each specified category.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter
Groups:
- Dupilumab 100mg q2w: Dupilumab 100 mg (in 0.67 mL for <=30 kg BW), SC injection q2w for 52 weeks in combination with stable-dose background therapy of medium-dose ICS with a second controller medication (i.e., LABA, LAMA, LTRA or methylxanthines) or high-dose ICS alone or high-dose ICS with second controller medication. Albuterol/salbutamol or levalbuterol/levosalbutamol was given as reliever medication. Participants were followed up for 12 weeks after last dose (i.e. up to Week 64).
- Dupilumab 200mg q2w: Dupilumab 200 mg (in 1.14 mL for >30 kg BW), SC injection q2w for 52 weeks in combination with stable-dose background therapy of medium-dose ICS with a second controller medication (i.e., LABA, LAMA, LTRA or methylxanthines) or high-dose ICS alone or high-dose ICS with second controller medication. Albuterol/salbutamol or levalbuterol/levosalbutamol was given as reliever medication. Participants were followed up for 12 weeks after last dose (i.e. up to Week 64).
Arm/Group | Dupilumab 100mg q2w | Dupilumab 200mg q2w
Number analyzed (Participants) | 91 | 179
nanograms per milliliter
  Baseline: number analyzed (Participants) | 90 | 178
  Baseline | 0.00 (948.683) | 0.00 (0.000)
  Week 6: number analyzed (Participants) | 87 | 172
  Week 6 | 28566.81 (47.114) | 50269.81 (46.667)
  Week 12: number analyzed (Participants) | 90 | 174
  Week 12 | 37741.97 (46.516) | 63476.17 (44.444)
  Week 24: number analyzed (Participants) | 90 | 173
  Week 24 | 42283.09 (47.910) | 49525.35 (52.806)
  Week 52: number analyzed (Participants) | 86 | 171
  Week 52 | 41467.97 (49.368) | 45295.35 (56.990)
  Week 64: number analyzed (Participants) | 4 | 15
  Week 64 | 39.00 (0.000) | 39.00 (0.000)

49. Secondary Outcome: Percentage of Participants With Treatment Emergent Antidrug Antibodies (ADA) Response
Description: ADA response was categorized as: treatment emergent and treatment boosted response. 1) Treatment emergent was defined as an ADA positive response in the assay post first dose, when baseline results were negative or missing. 2) Treatment boosted was defined as: an ADA positive response in the assay post first dose that was greater-than or equal to 4-fold over baseline titer levels, when baseline results were positive. The criteria for positive was defined as "30 to > 10,000", where low titer (< 1,000); moderate (1,000 <= titer <= 10,000) and high titer (> 10,000).
Time Frame: From Baseline up to Week 64
Population: Analysis was performed on ADA population which consisted of all participants who actually received at least 1 dose or part of a dose of the IMP, analyzed according to the treatment actually received and had at least one non-missing ADA result (either ADA negative or ADA positive) in the ADA assay after the first dose of IMP. Data for this outcome measure was planned to be collected and analyzed separately for dupilumab 100 mg and 200 mg dose.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dupilumab 100mg q2w | Dupilumab 200mg q2w
Number analyzed (Participants) | 133 | 91 | 178
percentage of participants
  Treatment-emergent ADA | 3.0 | 4.4 | 7.3
  Treatment-boosted ADA | 0 | 0 | 0

50. Secondary Outcome: Percentage of Participants With Seroconversion
Description: Seroconversion was defined as a post-vaccination titer >=40 (1/dilution) for those with a pre-vaccination titer <10 (1/dilution), or a >= 4-fold increase in post-vaccination titer for those with a pre-vaccination titer >=10 (1/dilution).
Time Frame: From Baseline up to Week 64
Population: Analysis was performed on safety population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 134 | 271
percentage of participants | 62.5 | 79.6

ADVERSE EVENTS:
Time Frame: All AEs were collected from signature of the informed consent form up to end of post treatment period (i.e., up to Week 64) regardless of seriousness or relationship to IMP.
Description: Reported AEs were treatment emergent AEs that developed/worsened in grade or became serious during during 'TEAE period' (from the time of first dose of study drug to the end of post-treatment period [i.e., up to Week 64]). Analysis was performed on safety population.
Arm/Group | Placebo | Dupilumab
All-Cause Mortality (participants affected / at risk) | 0/134 | 0/271
Serious Adverse Events (participants affected / at risk) | 6/134 | 13/271
Other Adverse Events (participants affected / at risk) | 89/134 | 161/271
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=134) | Dupilumab (N=271)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Immune Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Vision Blurred (Eye disorders) | 0 (0) | 1 (1)
Allergy To Chemicals (Immune system disorders) | 0 (0) | 1 (1)
Anaphylactic Reaction (Immune system disorders) | 1 (1) | 0 (0)
Drug Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Milk Allergy (Immune system disorders) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal Viral Infection (Infections and infestations) | 1 (1) | 0 (0)
Lymphadenitis Viral (Infections and infestations) | 1 (1) | 0 (0)
Parainfluenzae Virus Infection (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Hand Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Partial Seizures (Nervous system disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=134) | Dupilumab (N=271)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 15 (15)
Injection Site Erythema (General disorders) | 13 (93) | 35 (153)
Injection Site Oedema (General disorders) | 7 (15) | 28 (72)
Bronchitis (Infections and infestations) | 14 (22) | 17 (21)
Influenza (Infections and infestations) | 12 (17) | 20 (22)
Nasopharyngitis (Infections and infestations) | 29 (45) | 50 (76)
Pharyngitis (Infections and infestations) | 14 (19) | 23 (27)
Sinusitis (Infections and infestations) | 7 (10) | 9 (11)
Upper Respiratory Tract Infection (Infections and infestations) | 18 (30) | 35 (59)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 13 (17) | 33 (41)
Headache (Nervous system disorders) | 10 (17) | 18 (29)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 15 (17)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 16 (19) | 16 (27)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2019-10-18): https://cdn.clinicaltrials.gov/large-docs/59/NCT02948959/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-14): https://cdn.clinicaltrials.gov/large-docs/59/NCT02948959/SAP_001.pdf